CLINICAL TRIAL: NCT06734130
Title: A Phase IIA Study of Adaptive Androgen Deprivation and Docetaxel in Metastatic Castration Sensitive Prostate Cancer
Brief Title: Adaptive Androgen Deprivation and Docetaxel in Metastatic Castration Sensitive Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23260
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration Sensitive Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide; Triptorelin Pamoate; relugolix; enzalutamide; apalutamide; darolutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive Androgen Deprivation and Docetaxel Treatment (Experimental): This study will consist of various visits: a screening visit, 1-3 visits during the screening standard of care treatment period and visits every 4 weeks during the adaptive therapy period.
  Interventions: Drug: Luteinizing Hormone-Releasing Hormone (LHRH) analog; Drug: Androgen Receptor Signal Inhibitor (ARSI); Drug: Docetaxel

INTERVENTIONS:
Drug: Luteinizing Hormone-Releasing Hormone (LHRH) analog — The choice of the standard of care LHRH analog will be at the discretion of the treating physician.
  Other Names: Degarelix; Leuprolide; Triptorelin; Relugolix
Drug: Androgen Receptor Signal Inhibitor (ARSI) — The choice of the standard of care ARSI will be at the discretion of the treating physician.
  Other Names: Enzalutamide; Apalutamide; Darolutamide
Drug: Docetaxel — Docetaxel will be given by IV infusion at 75mg/m2 once every 3 weeks.

SUMMARY:
This is a prospective single center phase IIa open label nonrandomized study, which aims to test the hypothesis that the duration of castration sensitive phase of stage IV prostate cancer can be prolonged with adaptive androgen deprivation therapy (ADT) and Docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer and the diagnosis can be established through either prostate biopsy or biopsy of a metastatic lesion.
* No androgen deprivation therapy (ADT) with LHRH analog for more than 4 weeks after the diagnosis of metastatic prostate cancer. Prior ADT in the non-metastatic setting is allowed if it was given > 2 years prior to the diagnosis of metastatic prostate cancer.
* Achieved >50% PSA decline and <4 ng/ml PSA after the run-in period.
* Adequate organ function with absolute neutrophil count > 1000/l, Hb > 10 g/dl, Platelet > 100,000/l, Creatinine and liver enzymes within 1.5 folds of upper limits of normal.
* No uncontrolled arrhythmia; patients with h/o myocardia infarction or history of congestive heart failure, need to have estimated left ventricle ejection fraction above 40% either on echocardiogram or MUGA scan within 6 months of study enrollment.
* ECOG performance status 0-1.
* Non-sterilized men who are sexually active with a female partner of childbearing potential treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 weeks after last dose of ARSI or docetaxel administration.
* Ability to understand and the willingness to sign a written informed consent document or have a legally authorized representative sign on the subject's behalf. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Prior treatments with TAK-700/Orteronel, abiraterone, apalutamide or enzalutamide.
* Surgical castration.
* Documented liver or brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel (including any drugs formulated with polysorbate 80), or LHRH analog (e.g., leuprolide, triptorelin, relugolix, degarelix)
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs.
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of LHRH analog, or previously diagnosed with another malignancy & have any evidence of residual disease. Patients with early-stage skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with delayed healing of wounds, ulcers, and/or bone fractures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Castration Sensitivity Rate | Up to 36 months
  Percentage of patients who remain castration sensitive at 36 months from initiation of LHRH analog for stage IV prostate cancer.

SECONDARY OUTCOMES:
On treatment PSA Progression Free Survival | Up to 36 months
  On treatment PSA progression free survival will be analyzed using the Kaplan-Meier method.
Radiographic Progression Free Survival | Up to 36 months
  Radiographic progression free survival will be analyzed using the Kaplan-Meier method.
Overall Survival | Up to 36 months
  Overall survival will be analyzed using the Kaplan-Meier method.
Patient Reported Outcome | Up to 36 months
  Patient reported outcome as measured by National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Prostate Cancer Symptom Index -17 items (NFPSI-17).

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Caner Center, Tampa, Florida, United States